CLINICAL TRIAL: NCT05139251
Title: Positive Parenting: Empowering Young Mothers Experiencing Homelessness With a History of Inter-personal Violence to Improve Parenting Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Doncy Eapen, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HSC-SN-21-0869
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Positive Parenting
Keywords: Positive parenting; Women experiencing homelessness; Inter-personal violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recovering from Intimate partner violence through Strengths and Empowerment (RISE) +ePALS (Experimental)
  Interventions: Other: Recovering from Intimate partner violence through Strengths and Empowerment (RISE); Other: ePALS

INTERVENTIONS:
Other: Recovering from Intimate partner violence through Strengths and Empowerment (RISE) — RISE intervention will be implemented for a period of 4 weeks at the beginning of the program. Four components/modules of the RISE intervention which includes a) education on health effects of violence, b) improving coping and self-care, c) enhancing social support, and d) addressing sexual violence will be used. Toward the beginning of each session the participant will complete a brief survey including a 10-item general self-efficacy scale to be graphed and discussed together to provide more immediate feedback to women about their progress, and at times, inform module selection. At the conclusion of each RISE session, women are asked to set a goal related to the topic in consultation with the clinician
Other: ePALS — Participants and their children will then receive 6 weekly sessions of ePALS. The ePALS sessions include rapport building, recognizing and understanding children's signals, contingently responding to signals, labeling objects and actions, learning book reading strategies, maintaining children's focus of attention, helping children with self-regulation, and language scaffolding techniques. Each parent will have a personal parenting coach who remotely supports their progress through the program.
  After a parent views a PALS coaching session, they will videotape themselves trying the strategy for that week with their child. Then their coach sets up a zoom call and together they talk about the PALS strategy and view the video. The coach facilitates parental appraisal of their behavior and discuss what they thought worked with their child and what they want to do differently.

SUMMARY:
The purpose of this study is to strengthen the skills and self-efficacy of women by addressing the social and emotional trauma that they have experienced from inter-personal violence (IPRV) and homelessness and to promote positive parenting strategies through Play and Learning Strategies (ePALS), an evidence based intervention.

ELIGIBILITY:
Inclusion Criteria:

* women's report of physical, sexual or psychological abuse from a partner/ family member/ acquaintance/ stranger within the last 24 months
* have at least one child under the age of 5 years old

Exclusion Criteria:

* non-English speaking
* physical presence of a male partner at the time of enrollment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Change in Women's parenting stress as assessed by the Parental Stress scale (PSS) | Baseline, 1 month post intervention, 3 months post intervention
  PSS is an 18-item questionnaire and the participants rate each item on a scale ranging from 1 ("strongly disagree") to 5 ("strongly agree"), a higher score indicating more stress
Change in social support as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v 2.0 Emotional Support | Baseline, 1 month post intervention, 3 months post intervention
  The PROMIS emotional support tool has 16 items and the participants respond each item using a 5-point rating scale from 1(never)-5(always) a higher score indicating more emotional support
Change in social support as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v 2.0 Informational Support | Baseline, 1 month post intervention, 3 months post intervention
  The PROMIS informational support is a 10 items and participants respond each item using a 5-point rating scale (Health Measures) anchored by 1(never)-5(always) with a higher score indicating a better outcome
Change in women's empowerment as assessed by the Personal Progress Scale-Revised (PPS-R) | Baseline, 1 month post intervention, 3 months post intervention
  PPS-R is a 28-item self-report measure on which participants rate the extent to which they agreed or disagreed with each item on a 7-point scale.
Change in self efficacy as assessed by the General Self- Efficacy Scale (GSE) | Baseline, 1 month post intervention, 3 months post intervention
  GSE is a 10 item scale. Participants respond to statements such as "I can solve most problems if I invest the necessary effort" on a 4-point Likert scale anchored by 1(not at all true)-4( exactly true),the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Change in parent satisfaction as assessed by the Parenting Sense of Competence Scale (PSOC) | Baseline, 1 month post intervention, 3 months post intervention
  The PSOC is a 17-item scale and each item is rated on a 6-point Likert scale anchored by 1(strongly disagree to 6( strongly agree).A higher score indicates a higher parenting sense of competency
Change in children's behavior as assessed by the Devereux Early Childhood Assessments (DECA)-Infant | Baseline, 1 month post intervention, 3 months post intervention
  DECA (Infant) is a 33 item questionnaire for parents about their infants (1mont-18 months) It is a 5 point behavior rating scale scored from never to very frequently which provides an assessment of within-child protective factors central to social and emotional health and resilience.
Change in children's behavior as assessed by the Devereux Early Childhood Assessments (DECA)-Toddler | Baseline, 1 month post intervention, 3 months post intervention
  DECA (Toddler) is a 36 item questionnaire. It is a 5 point behavior rating scale scored from never to very frequently which provides an assessment of within-child protective factors central to social and emotional health and resilience.
Change in children's behavior as assessed by the Devereux Early Childhood Assessments (DECA)-Preschoolers | Baseline, 1 month post intervention, 3 months post intervention
  DECA (preschoolers) is a 38 item questionnaire. It is a 5 point behavior rating scale scored from never to very frequently which provides an assessment of within-child protective factors central to social and emotional health and resilience.
Change in perceived parent child connectedness as assessed by the Mothers Object Relational Scale- Short Form (MORS- SF) and MORS- Child scale. | Baseline, 1 month post intervention, 3 months post intervention
  this is a 14 item scale and each item is scored from 0( never)-5(always)

CONTACTS AND LOCATIONS:
Overall Officials: Doncy Eapen, PhD, RN, FNP-BC, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No